CLINICAL TRIAL: NCT00183040
Title: Hormonal Regulators of Muscle and Metabolism in Aging
Brief Title: HORMA: Hormonal Regulators of Muscle and Metabolism in Aging
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: AG0045; R01AG018169-01 (NIH); USC GCRC Protocol #1030
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2009-06-02 (Estimated); Status verified 2009-05

CONDITIONS: Sarcopenia; Muscle Weakness; Frailty
Keywords: andropause; hormone therapy; HRT
MeSH Terms: conditions — Sarcopenia; Muscle Weakness; Frailty | interventions — Testosterone; Growth Hormone

INTERVENTIONS:
Drug: Topical testosterone
Drug: Recombinant human growth hormone

SUMMARY:
The purpose of this study is to determine the relationship of deficiencies in testosterone and growth hormone to loss of muscle mass (sarcopenia) and functional impairment during aging and whether there is an interaction of these two hormone systems in maintaining normal skeletal muscle mass and physical function.

DETAILED DESCRIPTION:
Elderly persons experience progressive loss of skeletal muscle mass, muscle strength, and functional capacity for activities of daily living. Aging is also associated with a loss of hormones believed to be related to muscle and strength, namely testosterone and growth hormone (GH). The hypothesis being tested is that both hormone systems regulate musculoskeletal protein mass and contractile fibers by different and complimentary mechanisms and that optimal levels of both testosterone and GH are necessary to maintain skeletal muscle mass, muscular strength and power, and full functional activities of daily living during the aging process.

This is a controlled, 16 week study to evaluate the independent effects and interaction of these two anabolic hormone systems in community dwelling elderly men 65-90 years of age who are hyposomatotropic (deficiency of growth hormone) with low eugonadal status (total testosterone of 150-550 ng/dL). The study will utilize a two tiered randomization in which 108 study participants will first be randomized to either the low or high eugonadal level of testosterone using a novel Leydig cell clamp method (GnRH (gonadotropin-releasing hormone) agonist plus topical testosterone supplementation) to achieve target levels of testosterone. Low gonadal status (150-550 ng/dL) will be maintained with 5 g daily doses of topical testosterone, whereas high gonadal status (650-950 ng/dL) will be achieved with 10 g daily doses. Within these two groups, participants will be randomized to receive placebo or one of two doses of rhGH (recombinant human growth hormone) therapy (0, 3.0, 5.0 mcg/kg/day) in a double blinded fashion.

ELIGIBILITY:
Inclusion Criteria:

* Men who are 65-90 years of age
* Total serum IGF-1 (insulin-like growth factor) in the lower tertile for adults (56-167 ug/dl)
* Total serum testosterone of 150-550 ng/dL

Exclusion Criteria:

* BMI (Body Mass Index) 35 kg/m2 or greater
* Weight instability (>3% change in prior 3 months)
* Daily intake of total kilocalories less than or equal to 0.8X the RDA and intake of protein between 0.8 and 1.4 g/kg/day inclusive
* Acute illness in the prior 30 days
* Resistance training (wt lifting) in the past 12 months
* Vigorous aerobic sports (Competing as a Master athlete in the prior 5 years; weekly swimming, racquet ball, cycling, tennis, in preceding 12 months)
* Use of an anabolic agent (androgen, androgen precursor, rhGH, etc) in the preceding 12 months
* Use of medications that might affect amino acid metabolism (e.g. beta-adrenergic blockers, beta-agonists, Ca2+ channel blockers, corticosteroids)
* Fasting sugar greater than or equal to 126 mg/dl or diabetes requiring Rx
* History of benign intracranial hypertension
* Heart failure, active angina, or myocardial infarction in the prior 6 months or history of aortic stenosis
* Uncontrolled hypothyroidism or hyperthyroidism
* Rheumatoid arthritis, cirrhosis or active hepatitis
* History of carpal tunnel syndrome
* Prior cancer other than squamous or basal cell carcinoma of the skin
* Sleep apnea or severe chronic lung disease
* Anticoagulation with heparin or coumadin
* Blood pressure not controlled with medication to <180/95 mm Hg
* Calculated creatinine clearance <50 cc/min
* Serum prostatic antigen >4.0 or American Urological Association score greater than or equal to 8
* Hematocrit greater than or equal 52%, or ALT >1.5X ULN
* Failure to pass a modified Bruce treadmill stress test
* Severe disability limiting strength or physical function testing
* Dementia or cognitive impairment affecting a subject's ability to provide informed consent

Ages: 65 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2002-09; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
measures of fractional synthetic rates of mixed and contractile (actin and myosin heavy chain [MHC]) skeletal muscle proteins and degradation of skeletal muscle (ubiquitin, and proteasome sub-units)
analysis of local regulators of skeletal muscle synthesis (e.g. IGF-1, IGFBP4, myostatin).

SECONDARY OUTCOMES:
change in skeletal muscle strength, muscle mass, power and fatigability (endurance), physical performance, and markers of safety.

CONTACTS AND LOCATIONS:
Overall Officials: Fred R. Sattler, MD, Principal Investigator — Keck School of Medicine, University of Southern California
Locations (2):
- United States (2):
  - Tufts University, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri

REFERENCES:
- [Background] Dutta C, Hadley EC, Lexell J. Sarcopenia and physical performance in old age: overview. Muscle Nerve Suppl. 1997;5:S5-9. No abstract available. PMID 9331374
- [Background] Hasten DL, Pak-Loduca J, Obert KA, Yarasheski KE. Resistance exercise acutely increases MHC and mixed muscle protein synthesis rates in 78-84 and 23-32 yr olds. Am J Physiol Endocrinol Metab. 2000 Apr;278(4):E620-6. doi: 10.1152/ajpendo.2000.278.4.E620. PMID 10751194
- [Background] Urban RJ, Bodenburg YH, Gilkison C, Foxworth J, Coggan AR, Wolfe RR, Ferrando A. Testosterone administration to elderly men increases skeletal muscle strength and protein synthesis. Am J Physiol. 1995 Nov;269(5 Pt 1):E820-6. doi: 10.1152/ajpendo.1995.269.5.E820. PMID 7491931
- [Background] Ferrando AA, Sheffield-Moore M, Yeckel CW, Gilkison C, Jiang J, Achacosa A, Lieberman SA, Tipton K, Wolfe RR, Urban RJ. Testosterone administration to older men improves muscle function: molecular and physiological mechanisms. Am J Physiol Endocrinol Metab. 2002 Mar;282(3):E601-7. doi: 10.1152/ajpendo.00362.2001. PMID 11832363
- [Background] Blackman MR, Sorkin JD, Munzer T, Bellantoni MF, Busby-Whitehead J, Stevens TE, Jayme J, O'Connor KG, Christmas C, Tobin JD, Stewart KJ, Cottrell E, St Clair C, Pabst KM, Harman SM. Growth hormone and sex steroid administration in healthy aged women and men: a randomized controlled trial. JAMA. 2002 Nov 13;288(18):2282-92. doi: 10.1001/jama.288.18.2282. PMID 12425705
- [Derived] Yarasheski KE, Castaneda-Sceppa C, He J, Kawakubo M, Bhasin S, Binder EF, Schroeder ET, Roubenoff R, Azen SP, Sattler FR. Whole-body and muscle protein metabolism are not affected by acute deviations from habitual protein intake in older men: the Hormonal Regulators of Muscle and Metabolism in Aging (HORMA) Study. Am J Clin Nutr. 2011 Jul;94(1):172-81. doi: 10.3945/ajcn.110.010959. Epub 2011 May 4. PMID 21543538